CLINICAL TRIAL: NCT05261607
Title: Epidemiological Analysis of the Evolution of the Case-mix and Mortality in the Intensive Care Unit of Hospital Universitario De Getafe (1991-2026)
Brief Title: Analysis of the Evolution of Mortality in an Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Fernando Frutos-Vivar, Principal Investigator, Hospital Universitario Getafe
Other Study IDs: Evolution mortality ICU
Record Dates: First submitted 2022-01-12; First posted 2022-03-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-03

CONDITIONS: Intensive Care Unit; Mortality; Epidemiology; Respiration, Artificial; Sepsis Syndrome; Respiratory Failure; Neurologic Disorder
Keywords: Intensive care units; Outcome; Mortality
MeSH Terms: conditions — Respiratory Aspiration; Systemic Inflammatory Response Syndrome; Respiratory Insufficiency; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The intensive care units is of the main components of modern healthcare systems. Formally, its aim is to offer the critically ill health care fit to their needs; ensuring that this health care is appropriate, sustainable, ethical and respectful of their autonomy. Intensive medicine is a cross-sectional specialty that encompasses a broad spectrum of pathologies in their most severe condition, and specifically has as its foundation the practice of comprehensive care of the patient with organ dysfunction and susceptible to recovery. Although critically ill patients are a heterogeneous population, they have in common the need for a high level of care, often requiring the use of high technology, specific procedures for the support of organ dysfunction and the collaboration of other medical and surgical specialties for their management and treatment.

Since their origins in the late 1950s, intensive care units have been adapting to the changes arising from the best scientific evidence. In the late 1990s and early 2000s, there were some successful clinical trials published that had tested alternative management strategies in the ICU.

Mechanical ventilation is an intervention that defines the critical care specialty. Between 1970 and the 1990s, the management focused on normalizing arterial blood gas with aggressive mechanical ventilation. Over the ensuing decades, it became apparent that performing positive pressure ventilation worsened lung injury. The pivotal moment in the mechanical ventilation story would be the low versus high tidal volume trial. This trial shifted the focus away from normalizing gas exchange to reducing harm with mechanical ventilation. Further, it paved way for further trials testing ventilation interventions (PEEP strategy, prone position ventilation) and nonventilation interventions (neuromuscular blockade, corticosteroids, inhaled nitric oxide, extracorporeal gas exchange) in critically ill patients.

That evidence-based intensive care medicine has undoubtedly had an influence on the outcome of critically ill patients, in general, and, particularly, of patients requiring mechanical ventilation. Temporal changes in mortality over the time have been scarcely reported for patients admitted to intensive care unit.

Objective of this study is to estimate the changes over the time in several outcomes in the patients admitted to an 18-beds medical-surgical intensive care unit from 1991 (year of start of activity) to 2026

ELIGIBILITY:
Inclusion Criteria:

• Patients admitted to intensive care unit

Exclusion Criteria:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who required a admission to intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 1991-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit Mortality | 180 days
  Died during stay in the intensive care unit

SECONDARY OUTCOMES:
Hospital Mortality | 180 days
  Died during stay in the hospital
Mortality 28-day | 28 days from date of admission in the Hospital
  Mortality at day 28 after admission in the Hospital
Use of Mechanical ventilation | 180 days
  Proportion of patients who required mechanical ventilation (invasive and non-invasive) during stay in the intensive care unit
Length of stay in the intensive care unit | 180 days
  Stay in the intensive care unit
Length of stay in the hospital | 180 days
  Stay in the hospital
Complications/events during stay in the intensive care unit | 180 days
  Rate of complications/events occurred in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Frutos-Vivar, MD, Principal Investigator — Hospital Universitario de Getafe
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided